CLINICAL TRIAL: NCT00006137
Title: Pilot Study of Enalapril and Renal Function in Patients With IgA Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Stanford University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15244; SUMC-GCRC-5R01DK49372
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-09

CONDITIONS: IGA Glomerulonephritis
Keywords: IgA glomerulonephritis; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Glomerulonephritis, IGA; Rare Diseases; Urogenital Diseases | interventions — Enalapril

INTERVENTIONS:
Drug: enalapril

SUMMARY:
OBJECTIVES: I. Determine the most sensitive outcome measures (functional or morphological) of a progressive renal injury in patients with IgA nephropathy.

II. Determine which of these patients are destined to progress to further injury in order to target them for therapy.

III. Elucidate the determinants of progression in those patients who exhibit evidence of either increasing impairment of ultrafiltration capacity or ongoing destruction of nephrons.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive oral enalapril daily. Treatment continues for 5 years in the absence of unacceptable toxicity.

Patients undergo renal function studies every 6-12 months for 5 years. Patients undergo renal biopsy at 36-48 months after study entry.

ELIGIBILITY:
Histologically confirmed IgA nephropathy, diagnosed within the past 3 years

Clinical presentation of either isolated hematuria/proteinuria for less than 3 years OR

Acute nephritic or nephrotic syndrome

No secondary forms of IgA nephropathy associated with chronic inflammatory disease of the bowel and liver

No end stage renal failure as defined by the following: Glomerular filtration rate less than 15 mL/min AND Extensive glomerulosclerosis and tubulointerstitial damage

No systemic lupus erythematosus or systemic (extrarenal) vasculitis (Henoch-Schonlein syndrome)

Healthy volunteers will be accrued as a control group

No other concurrent medical or psychiatric illness that would preclude study

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Bryan D. Myers, Study Chair — Stanford University